CLINICAL TRIAL: NCT02206711
Title: Pharmacokinetics and Metabolism of [14C] BMS-955176 in Healthy Male Subjects
Brief Title: Study of the Absorption, Metabolism, and Route of Elimination of a Novel Class of Anti-HIV 1 Drugs (BMS-955176) in Humans.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 206291; AI468-036 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — BMS-955176

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single oral dose of [14C] BMS 955176 (Experimental): A single 180 mg oral dose of [14C] BMS-955176 containing approximately 80 microcurie of total radioactivity.
  Interventions: Drug: BMS-955176
- Nasoduodenal (ND) Tube Cohort (Experimental): A single dose of [14C] BMS 955176 on Day 1 with ND placement 1 hour post dose to facilitate continuous bile collection though 8 hours post dose.
  Interventions: Drug: BMS-955176

INTERVENTIONS:
Drug: BMS-955176 — Single dose of drug on Day 1

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK), metabolism, routes and extent of elimination, safety and tolerability of a single oral dose of [14C] BMS-955176 in healthy male subjects. There is no formal research hypothesis to be statistically tested for this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male subjects
* Ages 18-50 years
* Body weight of at least 110 lbs (50kg)
* BMI of 18 to 32 kg/m^2
* non-smoking

Exclusion Criteria:

* Clinically significant diagnostic or therapeutic radiation exposure within the previous 12 months (eg serial X-ray or CAT scans, barium meals).
* gastrointestinal disease including gastrointestinal surgery
* constipation or irregular bowel movements

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-08-08 (Actual); Primary Completion 2014-09-09 (Actual); Study Completion 2014-09-09 (Actual)

PRIMARY OUTCOMES:
To asses the PK (AUC, Cmax) of a single oral dose | Day 1 through Day 13 (predose to 288 hours)
  Serial blood samples for PK parameters determined from plasma concentration versus time
To estimate extent of elimination of a single oral dose (% TRA recovery) | Day 1 through Day 13 (predose to 288 hours)
  Sample of urinary/fecal/bile will be collected for determining total recovery.

SECONDARY OUTCOMES:
Safety Assessment | Day 1 through Day 13
  Safety assessments based on review of adverse events, vital sign measurements, electrocardiograms, physical examinations, and clinical laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: Viiv Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Madison, Wisconsin, United States